CLINICAL TRIAL: NCT01168388
Title: Movement Disorder Survey in East China
Acronym: MDS
Status: Completed | Type: Observational
Sponsor: Sir Run Run Shaw Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Xingyue Hu, Sir Run Run Shaw Hospital
Other Study IDs: SirRRSH-001
Record Dates: First submitted 2010-07-21; First posted 2010-07-23 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2010-04

CONDITIONS: Primary Dystonia; Hemifacial Spasm
Keywords: Dystonia; Hemifacial spasm; Cervical dystonia; Blepharospasm
MeSH Terms: conditions — Dystonic Disorders; Hemifacial Spasm; Dystonia; Torticollis; Blepharospasm

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Movement disorder

SUMMARY:
Movement disorder involve recurring or constant muscle contractions causing squeezing or twisting movement, such as hemifacial spasm, blepharospasm, cervical dystonias etc. The most common focal dystonia was cervical dystonia in western countries according to previous studies, which is different from China in Chinese neurologists' opinion. And there is no such survey. So the investigators are conducting a movement disorder survey in east China to confirm it.

ELIGIBILITY:
Inclusion Criteria:

* Patients seeking treatment in movement disorder clinics(include naive or may have previously been to clinics)

Exclusion Criteria:

* Patients who have received this movement disorder survey

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients seeking treatment in movement disorder clinics in east China during April 2010 to August 2010.
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with primary dystonia | half year
  It is Cross-Sectional, service-based survey to study the primary dystonina prevalence in east China.

SECONDARY OUTCOMES:
Number of participants with hemifacial spasm | half year
  It is a Cross-Sectional survey to study the prevalence of hemifacial spasm in movement disorder of east China.
Number of participants with blepharospasm | half year
  It is a Cross-Sectional survey to study the prevalence of blepharospasm in movement disorder of east China.

CONTACTS AND LOCATIONS:
Overall Officials: Xingyue Hu, MD, Study Chair — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Castelon Konkiewitz E, Trender-Gerhard I, Kamm C, Warner T, Ben-Shlomo Y, Gasser T, Conrad B, Ceballos-Baumann AO. Service-based survey of dystonia in munich. Neuroepidemiology. 2002 Jul-Aug;21(4):202-6. doi: 10.1159/000059525. PMID 12065883
- [Background] Matsumoto S, Nishimura M, Shibasaki H, Kaji R. Epidemiology of primary dystonias in Japan: comparison with Western countries. Mov Disord. 2003 Oct;18(10):1196-8. doi: 10.1002/mds.10480. PMID 14534928
- [Background] Butler AG, Duffey PO, Hawthorne MR, Barnes MP. An epidemiologic survey of dystonia within the entire population of northeast England over the past nine years. Adv Neurol. 2004;94:95-9. No abstract available. PMID 14509660
- [Background] Muller J, Kiechl S, Wenning GK, Seppi K, Willeit J, Gasperi A, Wissel J, Gasser T, Poewe W. The prevalence of primary dystonia in the general community. Neurology. 2002 Sep 24;59(6):941-3. doi: 10.1212/01.wnl.0000026474.12594.0d. PMID 12297587
- [Background] Nutt JG, Muenter MD, Aronson A, Kurland LT, Melton LJ 3rd. Epidemiology of focal and generalized dystonia in Rochester, Minnesota. Mov Disord. 1988;3(3):188-94. doi: 10.1002/mds.870030302. PMID 3264051